CLINICAL TRIAL: NCT06433128
Title: Expanded Access to Fosmanogepix for Patients With Serious or Life-threatening Invasive Fungal Infections Who Have no Other Treatment Options
Brief Title: Expanded Access to Fosmanogepix for Patients With Serious or Life-threatening Invasive Fungal Infections
Status: Available | Type: Expanded Access
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP to Fosmanogepix
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Invasive Fungal Infections
Keywords: Fungal infection; Candida; Anti-fungal; Yeast; Mold; Rare mold
MeSH Terms: conditions — Invasive Fungal Infections; Mycoses; Torulopsis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Fosmanogepix solution for infusion — Fosmanogepix solution for infusion, 20 mg/mL for intravenous administration
Drug: Fosmanogepix 400 mg tablets — Fosmanogepix 400 mg tablets for oral administration

SUMMARY:
The EAP is intended to provide a treatment option for patients with proven or probable serious or life-threatening invasive fungal infection (in accordance with the EORTC-MSGERC criteria) who have exhausted their treatment options, primarily due to an infection with a resistant fungal pathogen, and for whom no other treatment options are available through marketed drugs or investigational agents in clinical studies ongoing in the respective indication.

ELIGIBILITY:
The EAP is intended to provide a treatment option for patients with proven or probable serious or life-threatening invasive fungal infection (in accordance with the EORTC-MSGERC criteria) who have exhausted their treatment options, primarily due to an infection with a resistant fungal pathogen, and for whom no other treatment options are available through marketed drugs or investigational agents in clinical studies ongoing in the respective indication.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult